CLINICAL TRIAL: NCT02601963
Title: A Randomized, Multicenter, Double-blind, Vehicle-controlled Study to Evaluate the Safety and Efficacy of Two Different Doses of a Topical Minocycline Foam Compared to Vehicle in the Treatment of Papulopustular Rosacea - Study FX2015-10
Brief Title: Safety and Efficacy Study of a Topical Minocycline Foam in Patients With Papulopustular Rosacea
Acronym: EMIRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study FX2015-10
Record Dates: First submitted 2015-10-19; First posted 2015-11-11 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Rosacea; Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FMX-103 1.5% (Experimental): The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied along with vehicle. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Interventions: Drug: FMX-103 1.5%
- FMX-103 3% (Experimental): The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied along with vehicle. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Interventions: Drug: FMX-103 3%
- Vehicle foam (0%) (Placebo Comparator): The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied along with vehicle. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Interventions: Drug: Vehicle foam (0%)

INTERVENTIONS:
Drug: FMX-103 1.5% — The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied compared to vehicle in patients with moderate-to-severe papulopustular rosacea. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Other Names: Minocycline foam 1.5%
  Arms: FMX-103 1.5%
Drug: FMX-103 3% — The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied compared to vehicle in patients with moderate-to-severe papulopustular rosacea. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Other Names: Minocycline foam 3%
  Arms: FMX-103 3%
Drug: Vehicle foam (0%) — The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied compared to vehicle in patients with moderate-to-severe papulopustular rosacea. The foam will be applied once daily to the face for the 12-week treatment duration of the study.
  Other Names: Placebo
  Arms: Vehicle foam (0%)

SUMMARY:
The purpose of this study is to see if the study drug, FMX-103, is safe to give and if it helps people with moderate-to-severe papulopustular rosacea.

The investigational product is FMX-103 minocycline foam. Two concentrations of the investigational product, 1.5% and 3%, will be studied along with vehicle. The foam will be applied once daily to the face for the 12-week treatment duration of the study.

Approximately 210 patients will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age is 18 years or older.
2. Participants have a moderate-to-severe rosacea excluding lesions involving the eyes and scalp.
3. Subject must have diagnosed rosacea for at least 6 months prior to screening.

Exclusion Criteria:

1. History of hypersensitivity or allergy to minocycline, any other tetracycline or any other component of the formulation such as Soybean oil or Coconut oil.
2. Women of child bearing potential who are pregnant, lactating (in the last 3 months) or planning to become pregnant during the study period.
3. Moderate or severe rhinophyma, dense telangiectasis (score 3, severe), or plaque- like facial edema.
4. Rosacea conglobata or fulminans, corticosteroid-induced rosacea or isolated pustulosis of the chin, facial erythrosis of known origin other than rosacea (e.g., known carcinoid syndrome).
5. Ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical ophthalmic or systemic antibiotics, papulopustular rosacea that requires medically indicated systemic treatment.
6. Bacterial folliculitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
the absolute change in inflammatory lesion count at Week 12 compared to Baseline. | Baseline to Week 12

SECONDARY OUTCOMES:
The dichotomized Investigator's Global Assessment (IGA) score at Week 12 compared to Baseline | Baseline to Week 12
Percent change in inflammatory lesion count at Week 12 compared to Baseline | Baseline to Week 12
The dichotomized modified Investigator's Global Assessment (mIGA) score at Week 12 compared to Baseline. | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mrowietz, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (16):
- Germany (16):
  - Berlin
  - Blaubeuren Abbey
  - Bochum
  - Buxtehude
  - Darmstadt
  - Dülmen
  - Düsseldorf
  - Friedrichshafen
  - Kiel
  - Mahlow
  - Mainz
  - Osnabrück
  - Schweinfurt
  - Selters
  - Stuttgart
  - Ulm

REFERENCES:
- [Derived] Mrowietz U, Kedem TH, Keynan R, Eini M, Tamarkin D, Rom D, Shirvan M. A Phase II, Randomized, Double-Blind Clinical Study Evaluating the Safety, Tolerability, and Efficacy of a Topical Minocycline Foam, FMX103, for the Treatment of Facial Papulopustular Rosacea. Am J Clin Dermatol. 2018 Jun;19(3):427-436. doi: 10.1007/s40257-017-0339-0. PMID 29396702